CLINICAL TRIAL: NCT02508220
Title: Short-term Effects of Oxytocin Nasal Spray on Chronic Tinnitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Berthold Langguth, MD, Ph.D. (Other)
Collaborators: Otosul -Otorrinolaringologia Sul-Fluminense (Unknown)
Responsible Party: Sponsor-Investigator, Berthold Langguth, MD, Ph.D., Chair of the Tinnitus centrum Regensburg, University of Regensburg
Organization: University of Regensburg (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Uni-Reg-Oxy-Tin
Record Dates: First submitted 2015-03-18; First posted 2015-07-24 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-07

CONDITIONS: Chronic Tinnitus
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oxy-Placebo (Other): Syntocinon first, Placebo second 2 puffs in each nostril
  Interventions: Drug: Syntocinon; Drug: Placebo
- Placebo-Oxy (Other): Placebo first, Syntocinon second 2 puffs in each nostril
  Interventions: Drug: Syntocinon; Drug: Placebo

INTERVENTIONS:
Drug: Syntocinon — Oxytocin nasal spray
  Other Names: Oxytocin
Drug: Placebo — distilled water in nasal spray
  Other Names: distilled water

SUMMARY:
The study compares the short-term tinnitus reduction following a single oxytocin intervention with a placebo control condition.

ELIGIBILITY:
Inclusion Criteria:

* chronic tinnitus with a duration > 6 months
* medical examination by an ENT specialist
* sufficient knowledge of the Portuguese language to follow the instructions and answer the questionnaires
* VAS score >4 points

Exclusion Criteria:

* vascular tinnitus
* muscular tinnitus
* conductive hearing loss
* previous experience with oxytocin nasal spray
* additional medications during the intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-07; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Change of tinnitus on VAS | 30 minutes after intervention
Change of Clinical global impression scale | 30 minutes after intervention

SECONDARY OUTCOMES:
Audiometry measured in dB HL | within one hour before intervention
  measured in dB HL
Minimum Masking Level measured in dB HL | within one hour before intervention
  measured in dB HL
Tinnitus Matching | within one hour before intervention
  Frequency measured in Hz